CLINICAL TRIAL: NCT02398669
Title: An Open-Label, Single Dose Study to Assess Pharmacokinetics, Safety and Tolerability of Lorcaserin Hydrochloride in Obese Pediatric Subjects 6 to 11 Years of Age
Brief Title: A Single Dose Pharmacokinetic Study of Lorcaserin Hydrochloride in Obese Pediatric Subjects 6 to 11 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APD356-A001-026
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Obesity
Keywords: Obesity; Lorcaserin hydrochloride; APD356; Pediatric; Pharmacokinetics
MeSH Terms: conditions — Obesity | interventions — lorcaserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lorcaserin 10 mg (Experimental): Cohort 1 - obese pediatric participants between age group of 6 and 8 years (inclusive) Cohort 2 - obese pediatric participants between age group of 9 and 11 years (inclusive)
  Interventions: Drug: Lorcaserin hydrochloride

INTERVENTIONS:
Drug: Lorcaserin hydrochloride — A single 10 mg dose of oral tablet formulation of lorcaserin hydrochloride will be administered with 240 mL of water.
  Other Names: APD356

SUMMARY:
Study will evaluate the pharmacokinetics (PK), safety and tolerability of a single 10 mg dose of lorcaserin hydrochloride in obese pediatric subjects 6 to 11 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 6 years to 11 years (up to 11 years and 364 days), inclusive, at Screening.
2. BMI greater than or equal to 99th percentile for age and gender as defined as:

   Age Boys Girls 6 21.6 23.0 7 23.6 24.6 8 25.6 26.4 9 27.6 28.2 10 29.3 29.9 11 30.7 31.5

   but less than or equal to 44kg/m2 at Screening.
3. Provide written informed consent signed by parent/legal guardian prior to entering the study or undergoing any study procedures. A written or verbal assent from the subjects will also be obtained.
4. Females aged at least 8 years should have a negative serum B-human chorionic gonadotropin (beta-hCG) at Visit 1 and a negative urine pregnancy test prior to receiving their first dose of study drug at Visit 2.
5. Willing and able to comply with all aspects of the protocol.
6. Able to swallow a single tablet.

Exclusion Criteria:

1. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical attention within 4 weeks of dosing
2. Evidence of disease that may influence the outcome of the study within 4 weeks of dosing (eg, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, cardiovascular system, or subjects who have a congenital abnormality in metabolism)
3. Secondary (chromosomal, endocrine, or metabolic) causes of obesity (eg, Prader-Willi syndrome, Down's Syndrome, untreated hypothyroidism, or Cushing's syndrome).
4. Any history of abdominal surgery that may affect PK evaluations (eg, hepatectomy, nephrotomy, digestive organ resection or any gastrointestinal procedure for the purpose of weight loss, which would slow gastric emptying).
5. Any clinically relevant symptom or organ impairment found by medical history, physical examinations, vital signs, electrocardiogram (ECG) finding, or laboratory test results that require medical treatment at Screening.
6. Special needs subjects who are unable to comprehend trial-related instructions (eg, mild to profound mental retardation, moderate to severe cognitive developmental delay, pervasive developmental disorders, autism).
7. Females who are sexually active.
8. Ongoing epilepsy or other seizure disorder, or use of medications for a seizure disorder within 6 months of the Screening or between Screening and Day 1.
9. History of congestive heart failure, pulmonary arterial hypertension, congenital heart disease, or organ transplantation.
10. Resting heart rate less than 50 or greater than 120 beats/min at Screening or predose on Day 1.
11. Systolic blood pressure (BP) greater than 140 mmHg or less than 90 mmHg or diastolic blood pressure greater than 90 mmHg or less than 60 mmHg at Screening or predose on Day 1.
12. Hypersensitivity to the study drug or any of its excipients.
13. Significant change in diet or level of physical activity within 1 month prior to dosing or change in weight of greater than 5 kg within 3 months prior to dosing.
14. Known to be human immunodeficiency virus (HIV) positive at Screening.
15. Active viral hepatitis (B or C) as demonstrated by positive serology at Screening.
16. Unable to attend scheduled visits (eg, lack of transportation) or lack of a parent/guardian to supervise study participation.
17. Enrolled in another clinical trial that involved pharmacotherapy, or medical device, within 30 days before informed consent.
18. Use of drugs with serotonergic activity within 4 weeks before dosing, including but not limited to selective serotonin-norepinephrine reuptake inhibitors (SNRIs), selective serotonin reuptake inhibitors (SSRIs), tricyclic antidepressants (TCAs), bupropion, triptans, and drugs that impair metabolism of serotonin (including monoamine oxidase inhibitors [MAOIs], linezolid), dextromethorphan, lithium, tramadol, antipsychotics or other dopamine antagonists.
19. Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect cytochrome P450 activities or transporters (eg, grapefruit, grapefruit juice, grapefruit containing beverages, apple or orange juice, vegetables from the mustard green family [eg, kale, broccoli, watercress, collard greens, kohlrabi, brussels sprouts, mustard] and charbroiled meats) is prohibited within 2 weeks before dosing.
20. Intake of herbal preparations containing St. John's Wort is prohibited within 4 weeks before dosing.
21. Treatment within 4 weeks of dosing with over-the-counter weight loss products or appetite suppressants (including herbal weight loss agents), or within 3 months of dosing with a prescription weight loss drug (eg, phentermine, sibutramine, orlistat) or lipid dissolving injections (eg, Lipodissolve).

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Plasma PK profile of lorcaserin and its primary metabolites (M1 and M5) | Day 1 at 1, 2, 3, 4, and 6 hours postdose, Day 2 (24 +/- 2 h postdose), Day 3 (48 +/- 2 h postdose), and Day 5 (96 +/- 2 h postdose)

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) / Serious Adverse Events (SAEs) as a measure of safety and tolerabilty | From signing of informed consent until 30 days from participant's last dose or until resolution
  Safety will be assessed by monitoring and recording all AEs and SAEs, monitoring hematology, blood chemistry and urine values, measuring vital signs and ECG, and the performing physical examinations.

CONTACTS AND LOCATIONS:
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States